CLINICAL TRIAL: NCT04646512
Title: Effects of Taurine Supplementation Associated With High Intensity Physical Training on Irisin Levels, Energy Expenditure and Body Composition of Obese Women
Brief Title: Taurine Supplementation and Exercise on Irisin Levels in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ellen Cristini de Freitas, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 51921115500005426
Record Dates: First submitted 2020-11-20; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Obesity
Keywords: Obesity; Exercise; Irisin; Taurine; Energy Expenditure
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: double blind trial
Who Masked: Participant, Investigator
Masking Description: Intervention with taurine and / or placebo supplementation and physical training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taurine group and exercise (Active Comparator): Intervention with taurine supplementation and physical training.
  Interventions: Dietary Supplement: Taurine group and exercise and placebo group and exercise; Other: Physical training with Deep Water Running
- Placebo group and exercise (Placebo Comparator): Intervention with placebo supplementation and physical training.
  Interventions: Dietary Supplement: Taurine group and exercise and placebo group and exercise; Other: Physical training with Deep Water Running

INTERVENTIONS:
Dietary Supplement: Taurine group and exercise and placebo group and exercise — Both groups supplemented with taurine and / or placebo will perform physical training.
Other: Physical training with Deep Water Running — There will be a physical training for eight weeks.

SUMMARY:
Irisin is a myocin secreted by skeletal muscle in stimulus to physical exercise and has been described as a possible therapeutic tool in the fight against obesity by triggering a cascade of signaling that triggers the expression of genes responsible for the increase in energy expenditure and browning of adipose tissue white cells by activating thermogenesis promoter mitochondrial proteins. Although the science is engaged in the search for evidences about the actions of the irisin, the physical exercise involved and the improvement in the levels of obesity, many mechanisms are still unknown. Since taurine by means of irisin-like pathways also increases energy expenditure, it is believed that taurine supplementation associated with high intensity aerobic physical exercise can optimize the effects of irisin, increasing energy expenditure and improving body composition in obesity.

DETAILED DESCRIPTION:
Introduction: Irisin is a myocin secreted by skeletal muscle when stimulated by physical exercise that promotes increased thermogenesis (browning effect). Similarly, taurine is also associated with modulations of energy metabolism with promising actions in the control of metabolic disorders. Thus, it is believed that chronic taurine supplementation associated with physical training can optimize irisin concentrations after exercise.

Objective: Evaluate the effects of taurine supplementation associated with interval aerobic training on plasma irisin concentrations, energy expenditure, body composition and physical fitness in obese women. Methods: Twenty-two women aged 25 to 45 years, sedentary, with grade I obesity (BMI ≥30-35 kg / m²) and without comorbidities will be recruited for the study. The subjects will be submited to a high intensity interval aerobic training for 8 weeks, being 3 times by week, for 50 minutes, associated to the supplementation with 3g of taurine or placebo.

Methods: Assessment of dietary intake, Resting Energy Expenditure (GER) by indirect calorimetry, body composition by deuterium oxide, anthropometric measurements, HPLC plasma analysis of taurine, multiplex irisin and physical fitness variables will be performed pre and post intervention. The results will be expressed as mean and standard deviation and the ANOVA test two way repeated measures mixed model will be applied, with post hoc Sidak, to verify differences and statistical interactions (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* This study included women with obesity grade I (BMI ≥30 - ≤35Kg/m²), sedentary, with no associated comorbidity, convenience sample.

Exclusion Criteria:

* Women classified as overweight, obesity grade II and grade III (morbid), who present comorbidities associated with obesity (pre-diabetes, diabetes, hypertension, dyslipidemia, cardiovascular diseases and diseases of bone metabolism); smokers; who use hormones, sports supplements and / or weight loss medications. Perform some type of nutritional monitoring followed by diet or weight loss guidelines and that have medical impediment to the practice of physical exercise.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Changes body weight | Two times: (1) First day and (2) 10 weeks after assessments, adaptation and intervention
  The body weight was measured by digital balance before and after the intervention
Changes body composition | Two times: (1) First day and (2) 10 weeks after assessments, adaptation and intervention
  The body composition was evaluated through deuterium oxide
Changes indirect calorimetry | Two times: (1) First day and (2) 10 weeks after assessments, adaptation and intervention
  With a gas analyzer (indirect calorimeter), we evaluated the metabolic rate and rest (REE) and oxidation of substrates (lipids and carbohydrates)
Changes in total cholesterol and lipid fractions | Two times: (1) First day and (2) 10 weeks after assessments, adaptation and intervention
  Collected in EDTA tubes, were centrifuged.
Changes in plasma taurine concentration | Two times: (1) First day and (2) 10 weeks after assessments, adaptation and intervention
  Collected in EDTA tubes, were centrifuged and the plasma taurine concentration was evaluated using HPLC (high performance liquid chromatography).
Changes in plasma irisin concentration | Two times: (1) First day and (2) 10 weeks after assessments, adaptation and intervention
  Collected in EDTA tubes, were centrifuged and the plasma irisin concentration was evaluated using Multiplex - Kit Human Myokine Magnetic Bead Panel.
Changes Food intake | Two times: (1) First day and (2) 10 weeks after assessments, adaptation and intervention
  Food registry of 3 days. The quantification of the daily intake of nutrients will still be made using sofware.
Changes in determination of lactate | Two times: (1) First day and (2) 10 weeks after assessments, adaptation and intervention
  Blood samples were collected by manual puncture of the earlobe in previously calibrated and heparinized capillary tubes, stored in eppendorf with sodium fluoride. Analyzed by electrochemical lactate analyser.
Changes Physical Performance | Two times: (1) First day and (2) 10 weeks after assessments, adaptation and intervention
  Maximum effort test, according to Wilder, Brennan e Schotte (1993).

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriela Batitucci, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No